CLINICAL TRIAL: NCT03313726
Title: The Effect of Androgen Deprivation Therapy on Prostate Specific Membrane Antigen (PSMA) in Prostate Cancer
Brief Title: The Effect of ADT on PSMA-PET.
Acronym: ADTPSMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: T83/2017
Record Dates: First submitted 2017-10-09; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer
Keywords: PSMA-PET
MeSH Terms: conditions — Prostatic Neoplasms | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GnRh-antagonist A (Experimental)
  Interventions: Drug: GnRH antagonist
- GnRh-antagonist B (Experimental)
  Interventions: Drug: GnRH antagonist

INTERVENTIONS:
Drug: GnRH antagonist — Administration of GnRh antagonist after baseline PSMA-PET at day 0 and then repeated PSMA-PET scans at day 7, day 14 and day 28 to define the timeframe of the SUV-max.
  Arms: GnRh-antagonist A
Drug: GnRH antagonist — Administration of GnRh-antagonist after baseline PSMA-PET at day 0 and then repeated scan at day in which SUV-max was observed in the Arm A (day 7, day 14 or day 28). Then robot assisted radical prostatectomy and lymphadenectomy are performed to verify the finding.
  Arms: GnRh-antagonist B

SUMMARY:
Phase A: To describe and to determine the maximum standardised uptake values (SUV) in prostate specific membrane antigen positron emission tomography (PSMA-PET) before ADT and 7, 14 and 28 days after ADT.

Phase B: To validate phase A results by comparing the PSMA-PET findings to histopathological analysis of regional lymph nodes acquired from radical prostatectomy specimens. PSMA-PET is done before ADT and at maximum SUV defined by the phase A.

DETAILED DESCRIPTION:
Positron emission tomography has been commonly and successfully used, in combination with CT and MRI devices, in the staging of intermediate or high risk prostate cancer. Proper staging is essential to guide the treatment options, which usually are radical prostatectomy or radiotherapy in localized prostate cancer or hormonal treatment in patients with metastasized disease, patients with hormonal relapse after radical radiotherapy or as an adjuvant treatment together with radiotherapy.

The use of PET imaging increases the sensitivity in the evaluation of lymph node involvement, as almost 80% of metastatic lymph nodes in prostate cancer are smaller than the threshold size usually measured with CT or MRI.

Nowadays new specific receptor targeted PET tracers in prostate cancer imaging has been introduced. One of the most used is 68Ga-PSMA that evaluates the expression of prostate-specific membrane antigen. This tracer has been rapidly taken into account for its better sensitivity and specificity in prostate cancer staging compared to the lipid metabolism tracers, like 11C/18F labeled fluorocholine or 11C-acetate.

In the recent literature it has been demonstrated for the first time on humans that PSMA expression, imaged with 68Ga-PSMA-11-PET, has increased in a patient with metastatic prostate cancer after androgen deprivation therapy (ADT).

These findings suggest that the use of hormonal therapy can affect the expression of PSMA and our hypothesis is that ADT therapy could increase the sensitivity of 68Ga-PSMA PET to detect nodal or distant metastasis in patients with prostate cancer. This prospective study consists in two phases. In phase A, 5 patients with newly diagnosed high risk prostate cancer with PSMA-positive nodal or distant metastasis screened by 68Ga-PSMA-11 PET/MRI, are given androgen deprivation therapy (ADT) with GNRH antagonist. After ADT therapy initiation, 68Ga-PSMA-11 PET/MRI is repeated at 7, 14 and 30 days to determine the highest PSMA expression based on SUVmax measurement.

In phase B, 20 high risk prostate cancer patients determined to undergo radical prostatectomy are screened with 68Ga-PSMA-11 PET/MRI, and then given GNRH antagonist therapy. 68Ga-PSMA-11 PET/MRI is repeated at the time of maximum PSMA expression based on phase A results. The patients then undergo radical prostatectomy and lymphadenectomy and imaging findings are matched with histological data.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 to 85 years old
* Language spoken: Finnish
* Diagnosis: Histologically confirmed adenocarcinoma of prostate
* Adequate histological sampling consisting of at least 3 biopsy samples from each lobe
* No previous surgical, radiation or endocrine treatment for prostate carcinoma
* Clinical stage: T1c-T4N0-2M0-1 (arm, A); T1c-T3NxMx (arm, B)
* Serum creatinine ≤ 1,5 x ULN
* Patient agrees to undergo surgery (arm, B)
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethical Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* Infections: Patient must not have an uncontrolled serious infection
* contraindications for MRI (cardiac pacemaker, intracranial clips etc)
* Prior usage of 5-ARI medication in past 12 months
* Patient preference for active surveillance as a method of prostate cancer management

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
GnRh-antagonist, A | 0, 7, 14 and 28 days after ADT initiation
  Maximum SUV in PSMA-PET
GnRh-antagonist, B | 0 and 7, 14 or 28 days after ADT initiation according to phase A
  Sensitivity and specificity of pre and post ADT 68Ga-PSMA-11 PET/MRI and standard clinical MRI using histology as a reference

SECONDARY OUTCOMES:
GnRh-antagonist, A | 0, 7, 14 and 28 days after ADT initiation
  Testosterone level (nmol/l)
GnRh-antagonist, A | 0, 7, 14 and 28 days after ADT initiation
  PSA level (ug/l)
GnRh-antagonist, B | 56 and 112 days after ADT initiation
  Testosterone level (nmol/l)
GnRh-antagonist, B | 56 and 112 days after ADT initiation
  EPIC-questionnaire total and hormonal score

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Ettala O, Malaspina S, Tuokkola T, Luoto P, Loyttyniemi E, Bostrom PJ, Kemppainen J. Prospective study on the effect of short-term androgen deprivation therapy on PSMA uptake evaluated with 68Ga-PSMA-11 PET/MRI in men with treatment-naive prostate cancer. Eur J Nucl Med Mol Imaging. 2020 Mar;47(3):665-673. doi: 10.1007/s00259-019-04635-7. Epub 2019 Dec 26. PMID 31879814